CLINICAL TRIAL: NCT05249023
Title: Mode of Action of Butyrate in the Human Colon
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Örebro University, Sweden (Other)
Responsible Party: Principal Investigator, Robert Brummer, Professor, Örebro University, Sweden
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Bolus
Record Dates: First submitted 2021-03-23; First posted 2022-02-21 (Actual); Last update posted 2022-02-21 (Actual); Status verified 2022-02

CONDITIONS: Irritable Bowel Syndrome (IBS); Healthy
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Irritable Bowel Syndrome (IBS) participants (Experimental): 100 mM sodium butyrate solution containing indigo carmine as a dye agent will be administered to subjects in this arm.
  Interventions: Other: Sodium butyrate bolus
- Healthy participants (Experimental): 100 mM sodium butyrate solution containing indigo carmine as a dye agent will be administered to subjects in this arm.
  Interventions: Other: Sodium butyrate bolus

INTERVENTIONS:
Other: Sodium butyrate bolus — On the test day participants suffering from IBS and healthy participants will undergo a distal colonoscopy procedure for the collection of mucosal biopsy specimens pre- and post-administration of a sodium butyrate solution (100 mM) at a selected area in the descending colon. Biopsies will be obtained from the colon pre- and 90 min post-administration of the intervention solution. Blood samples will be collected before and at six time-points after the intervention solution administration.

SUMMARY:
Butyrate has recently gained attention as an important microbial compound in human colon health. Several diseases, including Irritable Bowel Syndrome (IBS), have been linked with a loss of butyrate in the colon resulting in the hypothesis that butyrate is important for disease resistance. However, despite a plethora of preclinical evidence about butyrate's role in colon health, data from human studies are insufficient, largely due to the lack of available tools for colon-specific butyrate delivery and sampling. This project will elucidate butyrate's mode of action in the human colon and its implications for gut functioning in IBS and healthy participants by employing a unique in vivo human setting. Specifically, the regulatory capacity of butyrate on intestinal barrier function and the transcriptional host responses that are associated with an increase of butyrate in the colon will be determined. Moreover, butyrate's role as a signalling molecule for gut hormones and serotonin release will be studied.

ELIGIBILITY:
Inclusion Criteria:

* signed informed consent
* Fulfilled Rome IV diagnostic criteria for IBS (for IBS participants)

Exclusion Criteria:

* known gastrointestinal diseases
* previous complicated gastrointestinal surgery (including e.g. appendectomy or cholecystectomy)
* pregnancy or breast-feeding
* use of antibiotics within the last 12 weeks before the colonoscopy procedure
* regular consumption of probiotics within the last 4 weeks before the colonoscopy procedure
* use of laxatives or anti-diarrhoeals within the last 4 weeks before the colonoscopy procedure
* use of serotonin selective re-uptake inhibitors (SSRI) or serotonin nor-epinephrine re-uptake inhibitors (SNRI) with the last 12 weeks before the colonoscopy procedure
* alcohol or drug abuse
* latex allergy
* any other clinically significant disease/condition which in the investigator's opinion could interfere with the results of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2018-04-11 (Actual); Primary Completion 2021-02-19 (Actual); Study Completion 2021-02-19 (Actual)

PRIMARY OUTCOMES:
Colonic permeability ex vivo in Ussing chambers | Mucosal biopsies collected pre- and 90 min post-administration of the butyrate solution
  Difference in the translocation of FITC-labeled dextran and horseradish peroxidase between the study arms before and after exposure to the butyrate bolus

SECONDARY OUTCOMES:
Butyrate uptake ex vivo in Ussing chambers | Mucosal biopsies collected pre- and 90 min post-administration of the butyrate solution
  Difference in the uptake of C14-labelled butyrate between the study arms before and after exposure to the butyrate bolus
Regulation of gene expression | Mucosal biopsies collected pre- and 90 min post-administration of the butyrate solution
  Difference in the genome-wide transcriptional response to an increase of butyrate in the descending colon between the study arms before and after exposure to the butyrate bolus
Concentrations of blood glucagon like peptide-1 (GLP-1) | Blood samples collected before (0 min) and at six timepoints after the butyrate solution administration (5, 15, 30, 45, 60 and 90 min).
  Difference in blood levels of GLP-1 between the study arms before and after exposure to the butyrate bolus
Concentrations of blood glucagon like peptide-2 (GLP-2) | Blood samples collected before (0 min) and at six timepoints after the butyrate solution administration (5, 15, 30, 45, 60 and 90 min).
  Difference in blood levels of GLP-2 between the study arms before and after exposure to the butyrate bolus
Concentrations of blood peptide YY (PYY) | Blood samples collected before (0 min) and at six timepoints after the butyrate solution administration (5, 15, 30, 45, 60 and 90 min).
  Difference in blood levels of PYY between the study arms before and after exposure to the butyrate bolus
Concentrations of blood gastric inhibitory polypeptide (GIP) | Blood samples collected before (0 min) and at six timepoints after the butyrate solution administration (5, 15, 30, 45, 60 and 90 min).
  Difference in blood levels of GIP between the study arms before and after exposure to the butyrate bolus
Concentrations of blood insulin | Blood samples collected before (0 min) and at six timepoints after the butyrate solution administration (5, 15, 30, 45, 60 and 90 min).
  Difference in blood levels of insulin between the study arms before and after exposure to the butyrate bolus
Concentrations of blood glucagon | Blood samples collected before (0 min) and at six timepoints after the butyrate solution administration (5, 15, 30, 45, 60 and 90 min).
  Difference in blood levels of glucagon between the study arms before and after exposure to the butyrate bolus
Concentrations of blood leptin | Blood samples collected before (0 min) and at six timepoints after the butyrate solution administration (5, 15, 30, 45, 60 and 90 min).
  Difference in blood levels of leptin between the study arms before and after exposure to the butyrate bolus
Concentrations of blood glucose | Blood samples collected before (0 min) and at six timepoints after the butyrate solution administration (5, 15, 30, 45, 60 and 90 min).
  Difference in blood levels of glucose between the study arms before and after exposure to the butyrate bolus
Concentrations of blood serotonin | Blood samples collected before (0 min) and at six timepoints after the butyrate solution administration (5, 15, 30, 45, 60 and 90 min).
  Difference in blood levels of serotonin between the study arms before and after exposure to the butyrate bolus
Concentrations of blood metabolites in the gluconeogenic pathway | Blood samples collected before (0 min) and at six timepoints after the butyrate solution administration (5, 15, 30, 45, 60 and 90 min).
  Difference in blood levels of metabolites in the gluconeogenic pathway between the study arms before and after exposure to the butyrate bolus
Concentrations of blood butyrate | Blood samples collected before (0 min) and at six timepoints after the butyrate solution administration (5, 15, 30, 45, 60 and 90 min).
  Difference in blood levels of butyrate between the study arms before and after exposure to the butyrate bolus

OTHER OUTCOMES:
Gastrointestinal symptoms measured by Gastrointestinal Symptom Rating Scale-IBS | 1 week
  Difference in the frequency and severity of gastrointestinal symptoms between the study arms before and after the exposure to the butyrate bolus (13 items that measure the severity of IBS symptoms in five clusters (pain, bloating, constipation, diarrhea, and early satiety).
Food habits measured by an electronic food frequency questionnaire Mealq | 1 week
  Survey of participants food habits prior the exposure to the butyrate bolus.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Örebro, Örebro, Örebro County, Sweden

REFERENCES:
- [Derived] Scharf MW, Forsgard RA, Prado SBR, Ganda Mall JP, Repsilber D, Brummer RJ, Marques TM, Wall R. Acute effects of butyrate on intestinal permeability in patients with irritable bowel syndrome assessed by a novel colonoscopy research model. Gut Microbes. 2025 Dec;17(1):2545414. doi: 10.1080/19490976.2025.2545414. Epub 2025 Aug 14. PMID 40810534